CLINICAL TRIAL: NCT04428580
Title: Implementing Family-Based Treatment for Adolescent Anorexia Nervosa for Providers in Private Practice: A Feasibility Study
Brief Title: Implementing FBT for Adolescent AN for Providers in Private Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, James Dale Lock, Professor of Child Psychiatry and Pediatrics in the Department of Psychiatry and Behavioral Sciences and Director of the Eating Disorder Program for Children and Adolescents, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 56548; R34MH123596 (NIH)
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Online Training for Therapists
Keywords: FBT; Training; Fidelity; Anorexia; Anorexia Nervosa
MeSH Terms: conditions — Anorexia; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online Training (Experimental): 10 lectures that are self-paced with a maximum of three months to complete with each lecture bundle comprising of 5-8 short (about 4 minutes in length), didactic videos that discuss the treatment model and provide mock therapy session video clips (modeling FBT with a typical adolescent AN case), as well as supplementary readings and videotaped role-plays. Enrollees complete each lecture bundle and complete the assignments as they move through the training at their own pace, but to have completed all within the 3-month time frame. When the training is completed, therapists will proceed to schedule post-online supervision for a minimum of 1 case and a maximum of 2 cases over the course of 3 months.
  Interventions: Other: Online FBT Training
- Webinar Training (Active Comparator): 1-hour weekly webinar lectures that essentially is the FBT training that is conducted in person, just recorded. There will be lectures discussing the scientific evidence supporting FBT, how therapists set up treatment for FBT, main interventions used in FBT during each phase, and recorded role-plays illustrating interventions throughout the 3 phases. Enrollees watch each webinar video as it is released weekly over a 12 week (3 month period). When the training is completed, therapists will proceed to schedule post-online supervision for a minimum of 1 case and a maximum of 2 cases over the course of 3 months.
  Interventions: Other: Webinar FBT Training

INTERVENTIONS:
Other: Online FBT Training — Therapists will receive online training in Family-Based Treatment (FBT)
  Arms: Online Training
Other: Webinar FBT Training — Therapists will receive webinar training in Family-Based Treatment (FBT)
  Arms: Webinar Training

SUMMARY:
There is a critical need to disseminate efficacious psychosocial treatments for mental disorders as there is a significant gap between evidenced-based approaches and common clinical practice. One example of the need to improve dissemination and implementation of psychosocial treatments is for adolescent Anorexia Nervosa (AN), a serious mental disorder with an incidence rate of about 1% that can become life-threatening. Based on outcomes from a series of randomized clinical trials (RCTs), the first-line treatment for adolescent AN is Family-based Treatment (FBT); however, very few therapists are trained to use FBT for AN. Further, while approximately 45-50% of US mental health outpatient providers are in private practice, little attention has been paid to how best to train this group. Care for adolescent AN, in particular, is provided in private practice at high rates, because specialist programs in non-private settings are few and not readily accessible. Motivations, incentives, and rationale for learning evidence-based treatments (EBTs) differ in this group compared to therapists embedded in an organization or health care system. In this application, we propose to use an online training strategy to study the adoption of FBT to better understand factors that limit or enhance uptake and implementation of this treatment in private practice. We developed and piloted a self-directed enhanced online training (ET-FBT) aimed at improving therapist skills and knowledge related to key components of FBT for AN that predict patient outcome in a group of therapists of which 64% were in private practice. We propose to build on these findings to examine the feasibility of new methods to retain therapists during supervision, assess fidelity, and collect patient outcomes from clinicians in private practice. Thus, our specific aims are:

Aim 1: The overall aim of the study is to assess the feasibility of conducting a randomized clinical trial comparing two implementation strategies (online training vs webinar training) for training clinicians in private practice in FBT for AN. We predict that those randomized to online training will be retained, receive supervision, and provide patient data at higher rates than those who receive webinar training.

Aim 2: Patient outcomes (reflecting therapist effectiveness) will be assessed by comparing patient weight gain from session 1 to 4 of FBT before and after training (target for training effect) and compared between randomized groups. We predict a moderate efficacy signal difference favoring those who are received the online training. because of increased training in key components in the online training program.

Aim 3: Validate training effect by examining the association between therapist fidelity to FBT and patient outcomes. We predict that fidelity will be correlated (target validation) with patient outcome. The effects of therapeutic alliance, participation in supervision, and self-efficacy on both fidelity and patient outcome will be explored.

Aim 4: Explore BL factors associated with implementation processes (e.g. prior training, experience, family work).The primary significance of this study is its potential to increase the availability of FBT--the most effective treatment for adolescent AN. Increased availability of FBT will decrease cost, hospitalization, morbidity, mortality, and chronicity of the disorder.

ELIGIBILITY:
Inclusion Criteria:

* Therapists are eligible to participate if they have completed a masters or doctoral training in their field (psychology, psychiatry, family therapy, social work)
* Licensed in their respective state
* No reports of malpractice or loss of privileges at relevant clinical institutions
* Have computer/web access for online training and assessments
* No previous 2-day in-person workshop training in FBT
* Submit baseline data on fidelity rating and weight gain from week 1-4 from a previously treated adolescent with AN they have treated in the last 6 months or alternatively one that they treat within 3 months of the initial screening before starting the training.

Exclusion Criteria:

* Therapists who have had previous training in FBT are not eligible.
* Therapists who are unable to provide baseline data on fidelity rating and weight gain from week 1-4 from a previously treated adolescent with AN they have treated in the last 6 months or alternatively one that they treat within 3 months of the initial screening before starting the training will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Lock, MD, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Citron K, Johnson M, Matheson BE, Onipede ZA, Yang HJ, Bohon C, Le Grange D, Lock J. Study protocol for training providers in private practice in family-based treatment for adolescents with anorexia nervosa: A randomized controlled feasibility trial. Contemp Clin Trials. 2022 Sep;120:106889. doi: 10.1016/j.cct.2022.106889. Epub 2022 Aug 20. PMID 35998767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1143 participants started the online screening process and 426 completed screening. 393 who completed the screen had sufficient information included in screening in order to assess eligibility. 151 participants signed informed consent, 123 were randomized.
Groups:
- Online Training: Therapists receive enhanced online training in Family-Based Treatment (FBT)
- Webinar Training: Therapists will receive online webinar training in Family-Based Treatment (FBT)
Period: Overall Study
Arm/Group | Online Training | Webinar Training
Started | 61 | 62
Started Training | 61 | 62
Finished Training | 58 | 59
Started Clinical Case Consultation | 26 | 28
Completed Clinical Case Consultation | 20 | 27
Completed | 61 | 62
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Online Training | Webinar Training | Total
Number analyzed (Participants) | 61 | 62 | 123
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.4 (7.2) | 37.5 (10.1) | 36.9 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 61 | 119
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 54 | 57 | 111
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 55 | 57 | 112
  More than one race | 5 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 62 | 123

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment
Description: Number of recruited subjects who provide full baseline data set at a rate of 50%
Time Frame: 1 day (day of baseline assessment)
Measure: Count of Participants; unit: Participants
Arm/Group | Online Training | Webinar Training
Number analyzed (Participants) | 61 | 62
Participants | 61 | 62

2. Primary Outcome: Retention
Description: Number of recruited subjects who provide full post training data set at a rate of 50%
Time Frame: Week 12 (1 day at end of training)
Measure: Count of Participants; unit: Participants
Arm/Group | Online Training | Webinar Training
Number analyzed (Participants) | 61 | 62
Participants | 48 | 51

3. Secondary Outcome: Exploring Association Between Fidelity and Outcome
Description: A therapist fidelity questionnaire and reported patient weight outcomes (weight change from FBT session 1 to session 4).
Time Frame: Baseline and Follow-up (after supervision)
Measure: Count of Participants; unit: Participants
Arm/Group | Online Training | Webinar Training
Number analyzed (Participants) | 61 | 62
Participants | 7 | 9

ADVERSE EVENTS:
Time Frame: Average approximately 6 months (12 weeks of training plus up to 12 weeks for supervision)
Arm/Group | Online Training | Webinar Training
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/62
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/62
Other Adverse Events (participants affected / at risk) | 0/61 | 0/62

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04428580/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/80/NCT04428580/SAP_001.pdf
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/80/NCT04428580/ICF_002.pdf